CLINICAL TRIAL: NCT04828434
Title: Virtual CST - A Collaborative Proof of Concept Study With FaceCog HK in Response to the Covid-19 Pandemic
Brief Title: Virtual Individual Cognitive Stimulation Therapy: a Proof of Concept Study
Acronym: V-iCST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University College, London (Other)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17127/002/1
Record Dates: First submitted 2021-03-23; First posted 2021-04-02 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Dementia; Dementia, Vascular; Dementia, Mixed; Dementia With Lewy Bodies; Dementia Frontal; Dementia, Mild; Dementia Moderate; Dementia Alzheimers; Dementia of Alzheimer Type; Dementia, Multi-Infarct; Dementia Frontotemporal
Keywords: Dementia; Randomized Controlled Trial; Cognitive Stimulation; Mild to Moderate Dementia; Teletherapy; Psychosocial Interventions
MeSH Terms: conditions — Dementia; Dementia, Vascular; Mixed Dementias; Lewy Body Disease; Lymphoma, Follicular; Alzheimer Disease; Dementia, Multi-Infarct; Pick Disease of the Brain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single-blind. The assessor will be blinded. Due to the nature of the intervention, the facilitator, and participants cannot be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Individual Cognitive Stimulation Therapy (Experimental): Virtual Cognitive Stimulation Therapy (V-iCST), a psychosocial intervention, is a modified version of CST for people with mild to moderate dementia. Like the original CST, each of the 14 sessions will begin with a "warm-up activity," which includes an orientation task and discussion of current affairs, followed by a main activity.
  V-iCST will be prescribed to participants twice a week, for 7 weeks and each session is approx. 45 minutes. The intervention will be delivered by trained professionals, such as research staff, psychologists, and trainee clinical psychologists. All facilitators will have experience in dementia care and will have completed the CST training.
  Interventions: Other: Virtual Individual Cognitive Simulation Therapy
- Treatment as usual (No Intervention): Standard care.

INTERVENTIONS:
Other: Virtual Individual Cognitive Simulation Therapy — Virtual Individual Cognitive Stimulation Therapy (V-iCST) is an individual and virtual adaptation of Cognitive Stimulation Therapy (CST), a routine psychosocial treatment for people with mild to moderate dementia in the UK.
  Arms: Virtual Individual Cognitive Stimulation Therapy

SUMMARY:
Due to COVID-19, the routine treatment for dementia, Cognitive Stimulation Therapy (CST), is currently suspended in multiple countries. Access to treatment is, therefore, paramount. The investigators seek to bridge the current treatment gap with a virtual and individual form of CST, called Virtual Individual Cognitive Stimulation Therapy (V-iCST). This psychosocial intervention was adapted from the key principles of CST and developed within the Medical Research Council (MRC) framework for complex interventions. The investigators aim to evaluate the feasibility and acceptability of V-iCST in a Randomized Controlled Trial.

This is a feasibility randomized controlled trial (RCT) for Virtual Individual Cognitive Stimulation Therapy (V-iCST), an evidence-based teletherapy for people with mild to moderate dementia. This psychosocial intervention is adapted from a routine and established dementia treatment, Cognitive Stimulation Therapy, and developed within the Medical Research Council (MRC) framework for complex interventions.

DETAILED DESCRIPTION:
Dementia, a global epidemic, affects 50 million individuals worldwide. Cognitive Stimulation Therapy (CST) is the only non-pharmacological therapy recommended by the UK government to improve cognition for mild to moderate dementia. It is delivered in over 85% of National Health Services (NHS) services and is offered in 34 countries. Unfortunately, this routine treatment is suspended due to lockdown, even though people with dementia are disproportionately affected by COVID-19. Accessible treatment is a pressing need. Virtual Individual Cognitive Stimulation Therapy (V-iCST) aims to bridge this treatment gap as an evidence-based treatment for dementia, developed within the Medical Research Council (MRC) Framework for complex interventions using principles of CST. There may still be a demand for V-iCST post-pandemic because those with sensory impairments and lack of transport provision may prefer a virtual and individual treatment. The investigators aim to 1) design V-iCST; 2) evaluate V-iCST in a feasibility Randomized Controlled Trial (RCT). A sample of 34 participants will be recruited. Seventeen will be allocated to V-iCST, and 17 to treatment as usual (TAU), the control group. Data will be collected pre-and post-test. Dementia prevalence is projected to reach 152 million worldwide by 2050. Therefore, accessible treatment is paramount during the pandemic and beyond.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of dementia, according to the DSM-IV
2. MoCA - BLIND ≥ 2
3. Age ≥ 18
4. Ability to communicate in English
5. Ability to complete outcome measures
6. Capacity to consent
7. Consent to video-conferencing
8. Access to video-conferencing

Exclusion Criteria:

1) Illness and disability that affects participation (as deemed by researcher)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment (feasibility of V-iCST) | Descriptive data will be collected during the study and analysed post-intervention; through study completion, 2 years
  Feasibility of recruitment by successful recruitment of the target sample of 32 in a 24-month period.
Retention rate (feasibility of V-iCST) | Descriptive data will be collected during the study and analyzed post-intervention; at 9-week follow-up
  Retention rate of at least 75% of participants at 9-week follow-up.
Attendance and retention rate (acceptability of V-iCST) | Descriptive data will be collected during the study and analyzed post-intervention; at 9-week follow-up
  Overall attendance and retention rates among the participants (60%) at 9-week follow-up.
Negative of adverse events (acceptability of V-iCST) | Descriptive data will be collected during the study and analyzed post-intervention; through study completion, 2 years
  Any negative or adverse events related to the intervention
Fidelity (acceptability of V-iCST) | Descriptive data will be collected during the study and analyzed post-intervention; through study completion, 2 years
  Fidelity will also be assessed to ensure that facilitators adhered to the protocol. Fidelity will be evaluated by a) facilitators' completion of the fidelity checklist following each session; b) vide recordings of all sessions and an independent researcher rating fidelity with a random 10% of the recordings.

SECONDARY OUTCOMES:
Change in cognitive function | Pre-test (baseline: week 0) and post test (week 9)
  Exploratory outcome; measured pre-and post-intervention with Montreal Cognitive Assessment Blind Version (MoCA-BLIND) (Wittich et al., 2010). MoCA - BLIND is a short version of the Montreal Cognitive Assessment designed for the visually impaired. It consists of 6 items with scores from 0 to 22, where a low score indicates poor performance.
Change in cognitive function | Pre-test (baseline: week 0) and post test (week 9)
  Exploratory outcome; measured pre-and post-intervention with Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog) (Rosen et al., 1984). ADAS-Cog is a sensitive scale measuring cognitive function with more items on short-term memory. This scale is frequently used in dementia drug trials, and has 11 items, and a total score of 70, where the higher the score, the more severe the impairments.
Change in quality of life | Pre-test (baseline: week 0) and post test (week 9)
  Exploratory outcome; measured pre-and post-test with Quality of Life in Alzheimer's Disease (QoL-AD) (Logsdon et al., 2002). QoL-AD has 13-items, and a sum score range from 13 to 52; higher score denotes better quality of life.
Change in mood | Pre-test (baseline: week 0) and post test (week 9)
  Exploratory outcome; measured pre-and post-test with Geriatric Depression Scale (GDS), a dichotomous screening tool with 15 items. Participants answer "yes" or "no" to symptoms of depression. A score of 10 or higher indicates depression.
Change in communication | Pre-test (baseline: week 0) and post test (week 9)
  Exploratory outcome; measured pre-and post-test with Holden Communication Scale (Strom et al., 2016), a proxy-based instrument with 12 items developed to evaluate conversation, awareness, knowledge and communication. Each item contains five response options on a scale of 0 to 4, with a maximum score of 48. A higher score suggests difficulties with communication.
Change in engagement | Evaluated by an independent researcher through video recordings; up to 48 months.
  Exploratory outcome; measured with the Adapted Greater Cincinnati Chapter Well-Being Observation Tool (Adapted GCCWBOT) (Kinney & Rentz, 2005). An independent researcher will assess session recordings of every participant. Each evaluation will be 62 minutes, and 8 domains will be assessed: interest, attention, pleasure, self-esteem, normalcy, disengagement, sadness, and negative affect.

CONTACTS AND LOCATIONS:
Overall Officials: Aimee Spector, PhD, DClinPsy, Principal Investigator — UCL
Locations (1):
- UCL, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Study results will be published in peer-reviewed journals, doctoral theses and presented at conferences, and disseminated to the public through information sheets. Participants who indicate their interest in receiving further information regarding dissemination will be sent a letter with the main findings of the study upon completion.
Time Frame: Upon study completion.
Access Criteria: Email authors.

REFERENCES:
- [Background] Logsdon RG, Gibbons LE, McCurry SM, Teri L. Assessing quality of life in older adults with cognitive impairment. Psychosom Med. 2002 May-Jun;64(3):510-9. doi: 10.1097/00006842-200205000-00016. PMID 12021425
- [Background] Rosen WG, Mohs RC, Davis KL. A new rating scale for Alzheimer's disease. Am J Psychiatry. 1984 Nov;141(11):1356-64. doi: 10.1176/ajp.141.11.1356. PMID 6496779
- [Background] Kinney JM, Rentz CA. Observed well-being among individuals with dementia: Memories in the Making, an art program, versus other structured activity. Am J Alzheimers Dis Other Demen. 2005 Jul-Aug;20(4):220-7. doi: 10.1177/153331750502000406. PMID 16136845
- [Background] Holden UP, Woods RT. Positive approaches to dementia care. Edinburgh: Churchill Livingstone, 1995.
- [Background] Yesavage JA, Sheikh JI. Geriatric Depression Scale (GDS) Recent evidence and development of shorter version. Clin Gerontol. 1986;5(1-2):165-73.
- [Background] Wittich W, Phillips N, Nasreddine ZS, Chertkow H. Sensitivity and Specificity of the Montreal Cognitive Assessment Modified for Individuals who are Visually Impaired. Journal of Visual Impairment & Blindness. 2010;104(6):360-368.
- Available data/document: International Cognitive Stimulation Therapy Centre Website — http://www.ucl.ac.uk/international-cognitive-stimulation-therapy